CLINICAL TRIAL: NCT02473224
Title: Phase I Study to Determine the Optimal Human Dose for GII.2 Norovirus (Snow Mountain) Challenge Studies
Brief Title: Optimal Human Dose for GII.2 Norovirus (Snow Mountain) Challenge Studies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: 12-0034
Record Dates: First submitted 2015-06-04; First posted 2015-06-16 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-06-15

CONDITIONS: Gastroenteritis Norovirus
Keywords: challenge; GII.2; HID50; Norovirus; Snow Mountain filtrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Experimental): 9 secretor-positive subjects will receive 1.2x10^4 Genome Equivalent Copies (GEC) oral dose on Day 1; and 2 secretor-positive subjects will receive the placebo, n=11
  Interventions: Biological: Norovirus GII.2 Challenge; Other: Placebo
- Cohort 2 (Experimental): 9 secretor-positive subjects will receive either 1.2 x 10^2GEC, or 1.2 x10^6 GEC oral dose on Day 1, depending on the percentage of subjects with illness from Cohort 1; 2 secretor-positive subjects will receive the placebo, n=11
  Interventions: Biological: Norovirus GII.2 Challenge; Other: Placebo
- Cohort 3 (Experimental): 9 secretor-positive subjects will receive either 1GEC, 1.2 x 10^1 GEC, 1.2 x 10^2 GEC, 1.2 x 10^3 GEC, 1.2 x 10^5 GEC, 1.2 x 10^6 GEC, or 1.2 x 10^7 oral dose on Day 1, depending on the percentage of subjects with illness from Cohorts 1 and 2; 2 secretor-positive subjects will receive the placebo, n=11
  Interventions: Biological: Norovirus GII.2 Challenge; Other: Placebo
- Cohort 4 (Experimental): 8 secretor-negative and 3 secretor-positive subjects will receive 1.2 x 10^7 GEC oral dose on Day 1, n=11
  Interventions: Biological: Norovirus GII.2 Challenge; Other: Placebo

INTERVENTIONS:
Biological: Norovirus GII.2 Challenge — GII.2 Snow Mountain Norovirus Filtrate. Cohort 1: 1.2x10^4 Genome Equivalent Copies (GEC) oral dose on Day 1. Cohort 2: either 1.2 x 10^2 GEC or 1.2 x10^6 GEC oral dose on Day 1, depending on the results of prior Cohort 1. Cohort 3: either 1GEC, 1.2 x 10^1 GEC, 1.2 x 10^2 GEC, 1.2 x 10^3 GEC, 1.2 x 10^5 GEC, or 1.2 x 10^6 GEC, or 1.2 GEC x 10^7 oral dose on Day 1, depending on the percentage of subjects with illness from Cohorts 1 and 2. Cohort 4: optimal dose of GEC as determined by the results of cohorts 1-3
Other: Placebo — Placebo: 80 ml of sterile water for oral administration

SUMMARY:
This is a phase I, randomized, double blind, as well as partially blinded (for Cohort 4), placebo-controlled safety, illness, and infection study of a new experimental human challenge stock of the Norovirus genogroup II, genotype 2 (GII.2) isolate designated Snow Mountain virus (SMV). The study duration is 24 - 36 months. The primary objectives are to: 1) evaluate the safety and reactogenicity of the GII.2 Snow Mountain norovirus challenge stock and 2) determine a safe and optimal challenge dose of GII.2 Snow Mountain norovirus to achieve illness in a high proportion (= / > 75%) of subjects.

DETAILED DESCRIPTION:
This is a phase I, randomized, double blind, as well as partially blinded (for Cohort 4), placebo-controlled safety, illness, and infection study of a new experimental human challenge stock of the Norovirus genogroup II, genotype 2 (GII.2) isolate designated Snow Mountain virus (SMV), administered to healthy adults 18-49 years of age. Groups of 11 subjects each will be admitted to the inpatient hospital research unit, challenged with live SMV or placebo by oral administration, and remain in isolation in the unit for at least 4 days following challenge. The study duration is 24 - 36 months. Subjects will be followed post-challenge for safety, reactogenicity, and illness (primary objectives), and secondary or exploratory objectives including infection and immune responses. There will be multiple clinical assessments and collection of blood, emesis, saliva, and stool specimens. The primary objectives are to: 1) evaluate the safety and reactogenicity of the GII.2 Snow Mountain norovirus challenge stock and 2) determine a safe and optimal challenge dose of GII.2 Snow Mountain norovirus to achieve illness in a high proportion (= / > 75%) of subjects. The secondary objectives are to: 1) determine the rate of infection in study participants after norovirus GII.2 challenge, 2) determine the quantity and duration of virus shedding in stool by RT-qPCR, 3) estimate the median time to cessation of shedding, 4) determine the modified Vesikari score as a measure of gastroenteritis severity, 5) determine GII.2 Snow Mountain norovirus-specific Immunoglobulin titers by ELISA before and after the challenge, 6) determine the effect of pre-existing GII.2 Snow Mountain norovirus-specific immunoglobulin in serum and saliva on the rate of infection, 7) determine total and GII.2 Snow Mountain norovirus-specific IgA- and IgG-Secreting Cells in circulation by ELISpot assay, 8) once the optimal challenge dose is determined in secretor positive subjects: investigate the safety and illness rate using that dose of the GII.2 challenge stock in secretor negative subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject able to provide written informed consent
2. Male or non-pregnant females between the ages of 18 and 49 years, inclusive
3. Women of childbearing potential must be practicing abstinence or using an acceptable method of birth control for at least 30 days prior to enrollment through day 45 after receipt of the challenge virus. Male subjects must agree not to father a child prior to day 45 after receipt of the challenge virus

   * A woman is considered of childbearing potential unless post-menopausal (absence of menses for > /= 1 year) or surgically sterilized (tubal ligation, bilateral oophorectomy or hysterectomy)
   * Acceptable contraception methods for women include but are not limited to: sexual abstinence from intercourse with men, monogamous relationship with vasectomized partner who has been vasectomized for 6 months or more prior to the subject enrolling in the study, barrier methods such as condoms or diaphragms with spermicide or foam, effective devices (IUDs, NuvaRing) or licensed hormonal products such as implants, injectables or oral contraceptives
4. For women of childbearing potential, must have a negative serum or urine pregnancy test at screening and negative urine pregnancy test within 24 hours prior to challenge
5. Are in good general health, as determined by the study investigator within 60 days of challenge
6. Demonstrate knowledge and comprehension of the study by scoring >/= 70 percent on a quiz of the study protocol and policies
7. Willing and able to participate in all study visits, including an inpatient stay of at least 96 hours
8. Demonstrated to be H type I secretor positive for HBGA binding by assay of saliva (this applies to all cohorts except the SN cohort, which will include secretor negative subjects only)

Exclusion Criteria:

1. Have household contact with or have daily contact with children under 2 years of age or persons older than 70 years of age
2. Have expected occupational or social contact with immunocompromised individuals in the 8 weeks after challenge, including persons with HIV infection or active cancer, children <2 years of age, pregnant women or persons who are immunosuppressed (e.g. history of stem cell or organ transplantation). Individuals who provide any child day care services (in-home or non-residential facility) are also excluded
3. Are healthcare workers with patient contact in the 8 weeks after challenge
4. Are food service workers expected to prepare/handle food in the 8 weeks after challenge
5. Plan to be living in a confined environment (e.g. ship, camp, or dormitory) within 8 weeks after receiving the challenge strain
6. For females, are pregnant or plan to become pregnant at any time between the Screening Visit through 45 days after receipt of the challenge virus
7. Are breastfeeding or plan to breastfeed at any given time throughout the study
8. Have a history of gastroenteritis in the 4 weeks prior to challenge or any history of chronic or recurrent diarrhea or vomiting
9. Have a history of malabsorption or maldigestion disorder (e.g. celiac sprue), major gastrointestinal (GI) surgery, irritable bowel syndrome or any other chronic GI disorders that would interfere with the study, including chronic constipation or increased stool frequency
10. Have moderate or severe illness and/or an oral temperature >/=100.4 degrees F and/or diarrhea or vomiting within seven days prior to challenge
11. Have a pulse rate less than 55 beats per minute (bpm) or greater than 100 bpm. If heart rate is <55 bpm and the investigator determines that this is not clinically significant (e.g., athletes) and heart rate increases > 55 bpm on moderate exercise (two flights of stairs), subject will not be excluded
12. Have a systolic blood pressure less than 90 mmHg or greater than 140 mmHg on two separate measurements (screening and pre-challenge)
13. Have a diastolic blood pressure less than 50 mmHg or greater than 90 mmHg on two separate measurements (screening and pre-challenge)
14. Have long-term use (> /= 2 weeks) of high-dose oral (>/= 20 mg per day prednisone or equivalent) or parenteral glucocorticoids, or high-dose inhaled steroids for greater than 7 days in the last 6 months
15. Have an autoimmune, inflammatory, vasculitic or rheumatic disease, including but not limited to systemic lupus erythematosus, polymyalgia rheumatic, rheumatoid arthritis or scleroderma
16. Have HIV, hepatitis B, hepatitis C infection or untreated latent syphilis
17. Have a seizure disorder
18. Have an active malignancy, history of malignancy (excluding nonmelanotic skin cancer in remission without treatment for more than 5 years) or current use of immunosuppressive or cytotoxic therapy
19. Have positive fecal culture for E. coli O157:H7, Salmonella, Campylobacter, Yersinia, or Shigella, evidence of norovirus in the stool by RT-qPCR or pathogenic ova and parasites detected on microscopic examination at screening
20. Have abnormal screening laboratory test results per laboratory reported normal values for white blood cells (WBCs), hemoglobin (Hgb), platelets, absolute neutrophil count (ANC), elevated total bilirubin, potassium, sodium and hemoglobin A1c (HbA1c) and urine protein
21. Have a serum creatinine greater than 1.1 x ULN
22. Have an ALT (SGPT) greater than 1.1 x ULN
23. Have a chronic condition that the study physician feels would pose a threat to participating subjects, including, but not limited to solid organ or stem cell transplantation, diabetes, clinically significant history of immunosuppressive illness, gall bladder disease, heart disease, lung disease, pancreatic disease, renal disease or neurological disease 24. Have abnormal findings on screening electrocardiogram deemed clinically significant by study physician

25. Have ongoing drug abuse/dependence (including alcohol), or a history of these issues within 5 years of enrollment 26. Have a positive urine test for opiates 27. Have any medical, psychiatric, occupational, or behavioral problems that make it unlikely for the subject to comply with the protocol as determined by the investigator 28. Are unwilling to comply with study procedures including abstaining from smoking for the duration of the inpatient portion of the study 29. Have participated in a previous NoV challenge study or NoV vaccine study 30. Have received experimental products within 30 days before study entry or plan to receive experimental products at any time during the study 31. Plans to enroll in another clinical trial that could interfere with safety assessment of the investigational product at any time during the study period, including study interventions such as drugs, biologics or devices 32. Plan to donate blood during the course of the study 33. Have received a live vaccine within 30 days before study entry or plan to receive a live vaccine prior to Day 30 of the study 34. Have received an inactivated vaccine within 14 days before study entry or plan to receive an inactivated vaccine prior to Day 14 of the study 35. Have received parenteral immunoglobulin or blood products within 3 months of the study start, or plan to receive parenteral immunoglobulin or blood products within 3 months after receiving the study agent 36. Use of antibiotics within 7 days prior to entry into the inpatient facility 37. Use of any H2 receptor antagonists (e.g., Tagamet, Zantac, and Pepcid), proton pump inhibitors (e.g., Prilosec, Protonix, and Prevacid), or prescription acid suppression medication or over-the-counter (OTC) antacids in the 72 hours prior to NoV challenge 38. Use of prescription and OTC medications containing acetaminophen, aspirin, ibuprofen, and other non-steroidal anti-inflammatory drugs within 48 hours prior to NoV challenge 39. Regular use of laxatives or anti-motility agents 40. Have a history of allergy to sodium bicarbonate 40. Have a history of allergy to sodium bicarbonate

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Infectious Dose-50 based on infection rate after challenge with various doses | Day 2 to Day 5
Number of serious adverse events related to virus challenge | Day 1 to Day 180
Number of subjects experiencing any mild reactogenicity outcomes | Day 1 to Day 10
Number of subjects experiencing any moderate reactogenicity outcomes | Day 1 to Day 10
Number of subjects experiencing any severe reactogenicity outcomes | Day 1 to Day 10
Number of subjects experiencing Grade 3 adverse events | Day 1 to Day 30
Proportion of subjects with GII.2 Snow Mountain norovirus-associated illness following GII.2 challenge | Day 1 to Day 5

SECONDARY OUTCOMES:
Duration of diarrhea related to the challenge strain | Day 1 to Day 5
Duration of virus shedding in PCR-positive stool for each challenge dose | Day -60 to Day 75
Duration of vomiting related to the challenge strain | Day 1 to Day 5
Levels of pre-existing serum blockage IgG prior to challenge | Inpatient Admission
Levels of pre-existing serum IgA prior to challenge | Inpatient Admission
Levels of pre-existing serum IgG prior to challenge | Inpatient Admission
Levels of pre-existing serum salivary IgA prior to challenge | Inpatient Admission
Magnitude of virus shedding in PCR-positive stools, reported as GEC/ml | Day -60 to Day 75
Proportion of subjects excreting challenge virus in stool | Day 1 to Day 30
Proportion of subjects showing a >/= 4 fold rise in virus-specific serum IgG | Day 1 to Day 30
Proportion of subjects with =/> 4 fold rise in virus-specific salivary IgA | Day 1 to Day 45
Proportion of subjects with =/> 4 fold rise in virus-specific serum blockage IgG | Day 1 to Day 45
Proportion of subjects with =/> 4 fold rise in virus-specific serum IgG | Day 1 to Day 45
Proportion of subjects with >/= 4 fold rise in virus-specific serum IgA | Day 1 to Day 45
Proportion of subjects with norovirus specific IgA-ASC/10^6 PBMC (freshly isolated PBMCs) | Day 1 to Day 45
Proportion of subjects with norovirus specific IgG-ASC/10^6 PBMC (freshly isolated PBMCs) | Day 1 to Day 45
Severity of diarrhea related to the challenge strain, determined using the Vesikari Score | Day 1 to Day 5
Severity of vomiting related to the challenge strain, determined using the Vesikari Score | Day 1 to Day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Emory Vaccine Center - The Hope Clinic, Decatur, Georgia, United States

REFERENCES:
- [Derived] Rouphael N, Beck A, Kirby AE, Liu P, Natrajan MS, Lai L, Phadke V, Winston J, Raabe V, Collins MH, Girmay T, Alvarez A, Beydoun N, Karmali V, Altieri-Rivera J, Lindesmith LC, Anderson EJ, Wang Y, El-Khorazaty J, Petrie C, Baric RS, Baqar S, Moe CL, Mulligan MJ. Dose-Response of a Norovirus GII.2 Controlled Human Challenge Model Inoculum. J Infect Dis. 2022 Nov 11;226(10):1771-1780. doi: 10.1093/infdis/jiac045. PMID 35137154